CLINICAL TRIAL: NCT00301184
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of pGA2/JS7 DNA Vaccine and Recombinant Modified Vaccinia Ankara/HIV62 Vaccine in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Safety of and Immune Response to a DNA HIV Vaccine (pGA2/JS7) Boosted With a Modified Vaccinia HIV Vaccine (MVA/HIV62) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 065; 10140 (Registry Identifier: DAIDS ES Registry Number); 5P01AI049364-05 (NIH)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; HIV DNA Vaccine; Modified Vaccinia Ankara Vaccine
MeSH Terms: conditions — HIV Infections | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1A (Experimental): One 0.3 mg dose of DNA HIV vaccine or placebo administered at study entry and Month 2, followed by one dose of 1x10^7 TCID50 MVA or placebo at Months 4 and 6
  Interventions: Biological: pGA2/JS7 DNA; Biological: Modified vaccinia Ankara/HIV62
- 1B (Experimental): One 3.0 mg dose of DNA HIV vaccine or placebo administered at study entry and Month 2, followed by one dose of 1x10^8 TCID50MVA or placebo administered at Months 4 and 6
  Interventions: Biological: pGA2/JS7 DNA; Biological: Modified vaccinia Ankara/HIV62
- 2A (Experimental): One MTD (determined in Part 1) of DNA HIV vaccine or placebo administered at study entry. One dose of placebo or MTD of MVA at Months 2 and 6
  Interventions: Biological: pGA2/JS7 DNA; Biological: Modified vaccinia Ankara/HIV62
- 2B (Experimental): One dose of placebo or MTD of MVA administered at study entry and Months 2 and 6
  Interventions: Biological: Modified vaccinia Ankara/HIV62

INTERVENTIONS:
Biological: pGA2/JS7 DNA — DNA Vaccine
  Arms: 1A; 1B; 2A
Biological: Modified vaccinia Ankara/HIV62 — Recombinant Modified Ankara Vaccine
  Other Names: MVA

SUMMARY:
The purpose of this study is to determine the safety of and immune response to a DNA HIV vaccine, pGA2/JS7, followed by a modified vaccinia (smallpox) HIV vaccine, MVA/HIV62, in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through a safe and effective vaccine that will prevent HIV infection. DNA vaccines are inexpensive to construct, easily produced in large quantities, and stable for long periods of time. Recombinant modified vaccinia Ankara vaccines have been shown to be safe in humans, and immunogenicity after administration of both vaccines has been encouraging. When used together, a more robust immunologic response was associated with DNA HIV vaccine administration followed by modified vaccinia vaccine administration, compared to using either DNA or vaccinia vaccine alone. This study will evaluate the safety and immunogenicity of an experimental DNA HIV vaccine prime, pGA/JS7, followed by a similarly structured modified vaccinia boost, MVA/HIV62, in HIV uninfected adults. Participants in this study will be recruited only in the United States.

This study will be divided into 2 parts. Each participant will be involved with their part of study for 1 year. Participants in Part 1 will be randomly assigned to one of two different vaccination groups. Group 1A participants will be randomly assigned to receive either placebo or 2 lower doses of the DNA HIV vaccine (DNA) at study entry and Month 2, followed by 2 lower doses of the modified vaccinia vaccine (MVA) at Months 4 and 6. Group 1B will not enroll until safety and immunogenicity data from Group 1A have been evaluated. Group 1B participants will receive either placebo or two higher doses of DNA at study entry and Month 2, followed by two higher doses of MVA at Months 4 and 6.

Enrollment into Part 2 will begin only after safety data from Part 1 are reviewed. In Part 2, participants will be randomly assigned to one of two different vaccination groups. Within each group, participants will be randomly assigned to receive some series of vaccines or placebo. Group 2A participants will receive either placebo or the maximum tolerated dose (MTD) from Part 1 of DNA at study entry and MTD of MVA at Months 2 and 6. Group 2B participants will receive MTD of MVA at study entry and Months 2 and 6.

There will be 12 study visits over 12 months for Groups 1 and 2. There will be 11 study visits over 12 months for Groups 3 and 4. Medication history, a physical exam, an interview, HIV and pregnancy prevention counseling, and adverse events reporting will occur at all visits. Blood and urine collection and an electrocardiogram (ECG) will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Has access to a participating HIV Vaccine Trials Unit (HVTU) and is willing to be followed for the duration of the study
* Understands vaccination procedure
* Willing to receive HIV test results
* Good general health
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Received HIV vaccines in prior HIV vaccine trial
* Received vaccinia vaccine. More information on this criterion can be found in the protocol.
* Recreational cocaine or methamphetamine use within 12 months prior to study entry
* Immunosuppressive medications within 168 days prior to first study vaccine administration. Participants who use corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for mild, uncomplicated dermatitis are not excluded.
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days (for influenza or pneumococcal vaccines) or 30 days (for allergy treatment with antigen injections) prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, or social condition that would interfere with the study. More information about this criterion can be found in the protocol.
* Any job-related responsibility that would interfere with the study
* Allergy to egg products
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* History of or known active cardiac disease. More information on this criterion can be found in the protocol.
* Electrocardiogram (ECG) with clinically significant findings OR features that would interfere with assessments for myocarditis or pericarditis. More information on this criterion can be found in the protocol.
* Two or more of the following cardiac risk factors: elevated blood cholesterol (defined as fasting low density lipoprotein [LDL] of greater than 160 mg/dl); first-degree relative (e.g., mother, father, brother, sister) who had coronary artery disease before the age of 50; current smoker; or body mass index (BMI) greater than 35
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants whose syphilis infection was fully treated at least 6 months prior to study entry are not excluded.
* Severe and unstable asthma
* Diabetes mellitus type 1 or 2
* Thyroid disease requiring treatment
* Serious angioedema within the past 2 years
* Uncontrolled hypertension OR systolic blood pressure (BP) of 150 mmHg or greater or diastolic BP of 100 mmHg or greater
* BMI greater than 40
* Bleeding disorder
* Cancer. If a participant has had surgery to remove the cancer and, in the opinion of the investigator, the cancer is not likely to recur during the study period, the participant is not excluded.
* Seizure disorder
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnancy or breastfeeding, or plans to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2006-04; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse and serious experiences) | Throughout study
Immunogenicity, as defined by the protocol | Throughout study
Social impacts (negative experiences or problems reported by the participants) | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goepfert, MD, Study Chair — University of Alabama at Birmingham; Christine Mhorag Hay, MD, Study Chair — University of Rochester
Locations (6):
- United States (6):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - Vanderbilt Vaccine CRS, Nashville, Tennessee

REFERENCES:
- [Background] Cebere I, Dorrell L, McShane H, Simmons A, McCormack S, Schmidt C, Smith C, Brooks M, Roberts JE, Darwin SC, Fast PE, Conlon C, Rowland-Jones S, McMichael AJ, Hanke T. Phase I clinical trial safety of DNA- and modified virus Ankara-vectored human immunodeficiency virus type 1 (HIV-1) vaccines administered alone and in a prime-boost regime to healthy HIV-1-uninfected volunteers. Vaccine. 2006 Jan 23;24(4):417-25. doi: 10.1016/j.vaccine.2005.08.041. Epub 2005 Aug 24. PMID 16176847
- [Background] Goonetilleke N, Moore S, Dally L, Winstone N, Cebere I, Mahmoud A, Pinheiro S, Gillespie G, Brown D, Loach V, Roberts J, Guimaraes-Walker A, Hayes P, Loughran K, Smith C, De Bont J, Verlinde C, Vooijs D, Schmidt C, Boaz M, Gilmour J, Fast P, Dorrell L, Hanke T, McMichael AJ. Induction of multifunctional human immunodeficiency virus type 1 (HIV-1)-specific T cells capable of proliferation in healthy subjects by using a prime-boost regimen of DNA- and modified vaccinia virus Ankara-vectored vaccines expressing HIV-1 Gag coupled to CD8+ T-cell epitopes. J Virol. 2006 May;80(10):4717-28. doi: 10.1128/JVI.80.10.4717-4728.2006. PMID 16641265
- [Background] Mwau M, Cebere I, Sutton J, Chikoti P, Winstone N, Wee EG, Beattie T, Chen YH, Dorrell L, McShane H, Schmidt C, Brooks M, Patel S, Roberts J, Conlon C, Rowland-Jones SL, Bwayo JJ, McMichael AJ, Hanke T. A human immunodeficiency virus 1 (HIV-1) clade A vaccine in clinical trials: stimulation of HIV-specific T-cell responses by DNA and recombinant modified vaccinia virus Ankara (MVA) vaccines in humans. J Gen Virol. 2004 Apr;85(Pt 4):911-919. doi: 10.1099/vir.0.19701-0. PMID 15039533
- [Background] Smith JM, Amara RR, Campbell D, Xu Y, Patel M, Sharma S, Butera ST, Ellenberger DL, Yi H, Chennareddi L, Herndon JG, Wyatt LS, Montefiori D, Moss B, McClure HM, Robinson HL. DNA/MVA vaccine for HIV type 1: effects of codon-optimization and the expression of aggregates or virus-like particles on the immunogenicity of the DNA prime. AIDS Res Hum Retroviruses. 2004 Dec;20(12):1335-47. doi: 10.1089/aid.2004.20.1335. PMID 15650426
- [Background] Sutter G, Staib C. Vaccinia vectors as candidate vaccines: the development of modified vaccinia virus Ankara for antigen delivery. Curr Drug Targets Infect Disord. 2003 Sep;3(3):263-71. doi: 10.2174/1568005033481123. PMID 14529359
- [Background] Goepfert PA, Elizaga ML, Sato A, Qin L, Cardinali M, Hay CM, Hural J, DeRosa SC, DeFawe OD, Tomaras GD, Montefiori DC, Xu Y, Lai L, Kalams SA, Baden LR, Frey SE, Blattner WA, Wyatt LS, Moss B, Robinson HL; National Institute of Allergy and Infectious Diseases HIV Vaccine Trials Network. Phase 1 safety and immunogenicity testing of DNA and recombinant modified vaccinia Ankara vaccines expressing HIV-1 virus-like particles. J Infect Dis. 2011 Mar 1;203(5):610-9. doi: 10.1093/infdis/jiq105. Epub 2011 Jan 31. PMID 21282192
- [Derived] Elizaga ML, Vasan S, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. PLoS One. 2013;8(1):e54407. doi: 10.1371/journal.pone.0054407. Epub 2013 Jan 17. PMID 23349878